CLINICAL TRIAL: NCT05338385
Title: Readiness Outcomes Affecting Return to Sport 2.0: An Intervention Feasibility & Pilot Study
Acronym: ROAR 2:Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Matthew Milewski, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00039872
Record Dates: First submitted 2022-03-07; First posted 2022-04-21 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: ACL Tear
Keywords: ACL tear; Mental Skills; Psychological Readiness
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will receive mental skills training in addition to receiving standard-of-care ACL reconstruction and follow-up care. The goal of mental skills training is to help athletes maximize performance, reach self-determined goals, and build confidence in their fields of play. Many of the same tools that benefit athletes in sport performance also translate to their injury experience. Mental conditioning helps athletes navigate the many ups and downs that accompany ACL injury and recovery. Athletes are taught techniques to maintain their sport mindset by capitalizing on motivation, consistency, and resilience. One-on-one sessions are athlete-centered, and are designed to encourage exploration and growth through tangible mental skills strategies.
  Interventions: Behavioral: Mental Skills Coaching

INTERVENTIONS:
Behavioral: Mental Skills Coaching — Participants will partake in a 1-hour pre-op initial intake, followed by five 30-min follow-up sessions at 2 weeks, 6 weeks, 3 months, 6 months and 9-months post-op. All sessions will be one-on-one with the same master's-level mental skills coach. At each session, the provider will allow time for participants to share their current injury experience to date (i.e. how they are doing, challenges they have encountered). Following this, participants will be introduced to a series of mental skills tools, including but not limited to mindset awareness, motivation, cognitive restructuring, goal setting, and objective performance assessment. Participants will be provided with handouts outlining the strategies addressed to help maintain consistency of mental skills engagement between sessions.

SUMMARY:
This study aims to determine the feasibility of implementing a mental skills training intervention for adolescent athletes who tear their ACL and undergo ACL reconstruction surgery alongside receiving standard-of-care clinical treatment. The study will also determine if the mental skills coaching program has any effect on the psychological readiness of patients to return to sport after undergoing surgery and postoperative recovery and rehabilitation. If feasible and if the mental skills training program shows promising effect on athletes' confidence in returning to sport, a large-scale clinical trial can be explored to assess the relationship between mental skills' impact on readiness to return to sport, which could in turn provide evidence on the benefits of integrating mental skills directly into standard clinical care.

DETAILED DESCRIPTION:
Approximately 350,000 individuals undergo anterior cruciate ligament (ACL) surgery with using allograft or autograft in the US annually. Even with successful ACL surgery, subsequent ACL tear occurs at a rate of 2-24% in physically active population. Most published reports focused on the young adult population, but few studies have focused on physically active young athletes and their return to sports (RTS) after surgery. As successful RTS following ACL reconstruction can be physically and psychologically challenging, increased attention has been directed to better understand the role a patient's psychological readiness to RTS plays in the rehabilitation phase, but there is an overall need to establish effective tools to help improve psychological readiness to RTS during this phase.

Mental skills training aims to improve athlete performance. Individuals involved in collegiate-level sports face the challenge of balancing rigorous athletic and academic demands. Given these demands, there is increasing need for programs to help athletes at varying levels and ages develop the skills necessary to maintain optimal performance. Such programs speak to the need for student-athletes to train their mental game much in the same way they train their physical game. They emphasize the value of and the ability to teach confidence, adaptability, and resilience.

Researchers have employed both mindfulness- and psychological skills-based techniques as means to promote student-athlete mental toughness and improved performance outcome. Mindfulness increases nonjudgmental awareness of the present, and is an effective treatment in non-sport related arenas. Psychological skills training educates athletes on how to improve strategies such as imagery, self-talk, goal setting, and arousal regulation. While these interventions may vary somewhat in terms of approach, there is evidence that both tactics positively impact athlete performance. We believe that these theories can be translated to athletes who are recovering from injuries and be used effectively to get patients back to their sports confidently.

The goal of mental skills training is to help athletes maximize performance, reach self-determined goals, and build confidence in their fields of play. Many of the same tools that benefit athletes in sport performance also translate to their injury experience. Mental conditioning helps athletes navigate the many ups and downs that accompany ACL injury and recovery. Athletes are taught techniques to maintain their sport mindset by capitalizing on motivation, consistency, and resilience. One-on-one sessions are athlete-centered, and are designed to encourage exploration and growth through tangible mental skills strategies. Topics that may be addressed include mindset awareness, goal setting, stress management, mental imagery, cognitive restructuring, and positive self-talk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a complete anterior cruciate ligament (ACL) tear
* Undergoing ACL reconstruction at Boston Children's Hospital by a study-participating surgeon
* Age at time of surgery between 8 and ≤ 25
* English-speaking

Exclusion Criteria:

* Torn medial collateral ligament (MCL), lateral collateral ligament (LCL), or posterior cruciate ligament (PCL) requiring reconstruction

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ACL-Return to Sports after Injury (ACL-RSI) | 6-9 months postop
  Questionnaire used to measure the psychological impact of returning to sport after ACL reconstruction surgery. Patients will complete this questionnaire at the clinic visit when they are cleared to RTS at either their 6-month or 9-month postoperative follow-up clinical visit. There are 12 questions that are rated on a 0-10 scale. Overall, this outcome measure is scored 0-100 (higher score = more psychologically ready to RTS). A score greater than or equal to 77% indicates that the patient is psychologically ready to RTS.
PROMIS Psychological Stress Experience - Bank (CAT version) | 6-9 months postop
  Assesses the thoughts or feelings about the world in the context of environmental or internal challenges. Patients will complete at the time of enrollment, any additional clinical visit, including 3 months, 6 months, and/or 9 months after surgery. There are 19 questions that are rated on a 1-5 scale. Overall, this outcome measure is scored 18-95 (lower score = less stress). Raw scores are then converted into T-scores.

OTHER OUTCOMES:
Compliance | Preop consult, 2 weeks postop, 6 weeks postop, 3 months postop, 6 months postop, 9 months postop
  Compliance will be calculated as the number of mental skills coaching sessions attended out of the six planned visits.
Proportion of Participation | Preop consult
  This will be defined as the number of people who agreed to participate in a mental skills course divided by the number of people who were approached.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Milewski, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wojtys EM, Brower AM. Anterior cruciate ligament injuries in the prepubescent and adolescent athlete: clinical and research considerations. J Athl Train. 2010 Sep-Oct;45(5):509-12. doi: 10.4085/1062-6050-45.5.509. No abstract available. PMID 20831399
- [Background] Hettrich CM, Dunn WR, Reinke EK; MOON Group; Spindler KP. The rate of subsequent surgery and predictors after anterior cruciate ligament reconstruction: two- and 6-year follow-up results from a multicenter cohort. Am J Sports Med. 2013 Jul;41(7):1534-40. doi: 10.1177/0363546513490277. Epub 2013 May 30. PMID 23722056
- [Background] Wright RW, Magnussen RA, Dunn WR, Spindler KP. Ipsilateral graft and contralateral ACL rupture at five years or more following ACL reconstruction: a systematic review. J Bone Joint Surg Am. 2011 Jun 15;93(12):1159-65. doi: 10.2106/JBJS.J.00898. PMID 21776554
- [Background] Paterno MV, Schmitt LC, Ford KR, Rauh MJ, Myer GD, Huang B, Hewett TE. Biomechanical measures during landing and postural stability predict second anterior cruciate ligament injury after anterior cruciate ligament reconstruction and return to sport. Am J Sports Med. 2010 Oct;38(10):1968-78. doi: 10.1177/0363546510376053. Epub 2010 Aug 11. PMID 20702858
- [Background] Oiestad BE, Holm I, Aune AK, Gunderson R, Myklebust G, Engebretsen L, Fosdahl MA, Risberg MA. Knee function and prevalence of knee osteoarthritis after anterior cruciate ligament reconstruction: a prospective study with 10 to 15 years of follow-up. Am J Sports Med. 2010 Nov;38(11):2201-10. doi: 10.1177/0363546510373876. Epub 2010 Aug 16. PMID 20713644
- [Background] Oiestad BE, Holm I, Engebretsen L, Risberg MA. The association between radiographic knee osteoarthritis and knee symptoms, function and quality of life 10-15 years after anterior cruciate ligament reconstruction. Br J Sports Med. 2011 Jun;45(7):583-8. doi: 10.1136/bjsm.2010.073130. Epub 2010 Jul 20. PMID 20647299
- [Background] Lohmander LS, Englund PM, Dahl LL, Roos EM. The long-term consequence of anterior cruciate ligament and meniscus injuries: osteoarthritis. Am J Sports Med. 2007 Oct;35(10):1756-69. doi: 10.1177/0363546507307396. Epub 2007 Aug 29. PMID 17761605
- [Background] Vealey, S. R. (2007). Mental skills training in sport. In G. Tenenbaum, R. Eklund, & R. Singer (Eds.), Handbook of sport psychology (pp. 287-309). Wiley. Hoboken, NJ.
- [Background] Humphrey, J. H., Yow, D. A., & Bowden, W. W. (2000). Stress in college athletics: Causes, consequences, coping. The Haworth Half-Court Press. Binghamton, NY.
- [Background] Kimball, A., & Freysinger, V. J. (2003). Leisure, stress, and coping: The sport participation of collegiate student-athletes. Leisure Sciences, 25(2-3), 115-141.
- [Background] Papanikolaou, Z., Nikolaidis, D., Patsiaouras, A., & Alexopoulos, P. (2003). The freshman experience: High stress-low grades. Athletic Insight: The On-line Journal of Sport Psychology, 5.
- [Background] Sallen J, Hemming K, Richartz A. Facilitating dual careers by improving resistance to chronic stress: effects of an intervention programme for elite student athletes. Eur J Sport Sci. 2018 Feb;18(1):112-122. doi: 10.1080/17461391.2017.1407363. Epub 2017 Dec 3. PMID 29199550
- [Background] Ajilchi B, Amini HR, Ardakani ZP, Zadeh MM, Kisely S. Applying mindfulness training to enhance the mental toughness and emotional intelligence of amateur basketball players. Australas Psychiatry. 2019 Jun;27(3):291-296. doi: 10.1177/1039856219828119. Epub 2019 Feb 14. PMID 30763131
- [Background] Jones BJ, Kaur S, Miller M, Spencer RMC. Mindfulness-Based Stress Reduction Benefits Psychological Well-Being, Sleep Quality, and Athletic Performance in Female Collegiate Rowers. Front Psychol. 2020 Sep 18;11:572980. doi: 10.3389/fpsyg.2020.572980. eCollection 2020. PMID 33071908
- [Background] Rothlin P, Birrer D, Horvath S, Grosse Holtforth M. Psychological skills training and a mindfulness-based intervention to enhance functional athletic performance: design of a randomized controlled trial using ambulatory assessment. BMC Psychol. 2016 Jul 26;4(1):39. doi: 10.1186/s40359-016-0147-y. PMID 27457721